CLINICAL TRIAL: NCT03003299
Title: A Prospective, Single-Arm, Multicenter Study to Investigate the Safety and Effectiveness of SAPIEN 3/SAPIEN 3 Ultra Transcatheter Heart Valve Implantation in Patients With a Failing Aortic Bioprosthetic Valve
Brief Title: PARTNER 3 Trial - Aortic Valve-in-Valve
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-08 AVIV
Record Dates: First submitted 2016-12-19; First posted 2016-12-28 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Aortic Stenosis; Aortic Stenosis, Severe
Keywords: SAPIEN 3; PARTNER 3; cardiovascular disease; heart disease; aortic stenosis; SAVR; TAVR; failing surgical valve; failing bioprosthetic valve; failing valve; SAPIEN 3 Ultra
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TAVR - Failing surgical or transcatheter valve (Experimental): Patients with a failing surgical or transcatheter bioprosthetic valve will undergo transcatheter aortic valve replacement (TAVR).
  Interventions: Device: Edwards SAPIEN 3/SAPIEN 3 Ultra THV

INTERVENTIONS:
Device: Edwards SAPIEN 3/SAPIEN 3 Ultra THV — Edwards SAPIEN 3/SAPIEN 3 Ultra THV system with the associated delivery systems.

SUMMARY:
This study will assess the safety and effectiveness of the SAPIEN 3/SAPIEN 3 Ultra transcatheter heart valve (THV) in patients with a failing aortic bioprosthetic valve.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multicenter study.

ELIGIBILITY:
Inclusion Criteria:

1. Failing surgical or transcatheter bioprosthetic valve in the aortic position demonstrating ≥ moderate stenosis and/or ≥ moderate insufficiency.
2. Bioprosthetic valve with a true internal diameter (True ID) of 18.5 mm to 28.5 mm.
3. NYHA Functional Class ≥ II.
4. Heart Team agrees the patient is low to intermediate risk.
5. Heart Team agrees valve implantation will likely benefit the patient.
6. The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Surgical or transcatheter valve in the mitral position (mitral rings are not an exclusion)
2. Severe regurgitation (> 3+) or stenosis of any other valve
3. Failing valve has moderate or severe paravalvular regurgitation
4. Failing valve is unstable, rocking, or not structurally intact
5. Increased risk of coronary obstruction by prosthetic leaflets of the failing valve.
6. Increased risk of embolization of THV
7. Known bioprosthetic valve with residual mean gradient > 20 mmHg at the end of the index procedure for implantation of the original valve
8. Iliofemoral vessel characteristics that would preclude safe placement of the introducer sheath (Transfemoral)
9. Anatomical characteristics that would preclude safe access to the ascending aorta (Transaortic)
10. Anatomical characteristics that would preclude safe access to the apex (Transapical)
11. Evidence of an acute myocardial infarction ≤ 30 days before enrollment
12. Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days prior to the index procedure. Implantation of a permanent pacemaker or implantable cardioverter defibrillator is not considered an exclusion.
13. Patients with planned concomitant surgical or transcatheter ablation for Atrial Fibrillation
14. Leukopenia, anemia, thrombocytopenia, history of bleeding diathesis or coagulopathy or hypercoagulable states
15. Untreated clinically significant coronary artery disease requiring revascularization
16. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation, or mechanical heart assistance within 30 days of enrollment
17. Emergency interventional/surgical procedures within 30 days prior to the procedure
18. Any planned surgical, percutaneous coronary, or peripheral procedure to be performed within the 30-day follow-up from the procedure
19. Hypertrophic cardiomyopathy with obstruction
20. LVEF < 30%
21. Cardiac imaging evidence of intracardiac mass, thrombus, or vegetation
22. Inability to tolerate or condition precluding treatment with antithrombotic/anticoagulation therapy during or after the valve implant procedure
23. Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with premedication
24. Stroke or transient ischemic attack within 90 days of enrollment
25. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 30 days of enrollment
26. Renal insufficiency and/or renal replacement therapy at the time of screening
27. Active bacterial endocarditis within 180 days of the procedure
28. Patient refuses blood products
29. Estimated life expectancy < 24 months
30. Positive urine or serum pregnancy test in female subjects of childbearing potential
31. Currently participating in an investigational drug or another device study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2017-01-05 (Actual); Primary Completion 2033-01 (Estimated); Study Completion 2038-04 (Estimated)

PRIMARY OUTCOMES:
Safety and Effectiveness - Non-hierarchical composite of all-cause mortality and stroke | 1 year
  Number of patients that died and/or had a stroke

SECONDARY OUTCOMES:
Mean gradient | 30 days
  Measures the mean aortic pressure gradient from the measured velocity. Units used are mmHg.
Peak gradient | 30 days
  Measures the peak aortic pressure gradient from the measured velocity. Units used are mmHg.
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 30 days
  Change from baseline in KCCQ. The KCCQ is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life.
New York Heart Association (NYHA) Classification | 30 days
  Change from baseline in NYHA. NYHA is a functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I - IV, with the lowest (I) as no limitations and the highest (IV) unable to carry on any physical activity without discomfort.
Six-Minute Walk Test (6MWT) | 30 days
  Change from baseline in 6MWT. The 6-Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Chris S Malaisrie, MD, Principal Investigator — Northwestern University Feinberg School of Medicine; Alan Zajarias, MD, Principal Investigator — Washington University School of Medicine; Mayra Guerrero, MD, Principal Investigator — Mayo Clinic
Locations (51):
- United States (50):
  - Banner University Medical Center, Phoenix, Arizona
  - University of California Los Angeles, Los Angeles, California
  - Sutter Medical Center, Sacramento, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - UC Health Northern Colorado/Medical Center of the Rockies, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - JFK Medical Center/ Atlantic Clinical Research Collaborative, Atlantis, Florida
  - University of Florida, Gainesville, Gainesville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Northshore University HealthSystem, Evanston, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City Mid America, Kansas City, Missouri
  - Washington University/ Barnes-Jewish Hospital, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Newark Beth Israel, Newark, New Jersey
  - University of Buffalo, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - New York University (NYU) Langone Medical Center, New York, New York
  - Cornell University, New York, New York
  - Columbia University Medical Center/ New York Presbyterian Hospital, New York, New York
  - Carolina's Health System, Charlotte, North Carolina
  - NC Heart and Vascular (Rex Hospital), Raleigh, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Providence Heart & Vascular Institute, Portland, Oregon
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Saint Thomas Health Services, Nashville, Tennessee
  - Austin Heart, PLLC, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - The Heart Hospital Baylor Plano, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Heart and vascular Instritute (Fairfax Inova), Fairfax, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - University of Wisconsin - Madison, Madison, Wisconsin
- St. Paul's Hospital, Providence Health Care, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No